CLINICAL TRIAL: NCT03755960
Title: Acupuncture in Symptomatic Diabetic Peripheral Neuropathy.
Brief Title: ACUpuncture in Diabetic Peripheral Neuropathy
Acronym: ACUDPN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benno Brinkhaus (Other)
Collaborators: Karl and Veronica Carstens Foundation (Other)
Responsible Party: Sponsor-Investigator, Benno Brinkhaus, Principal Investigator, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACUDPN; 1/183/18 (Other: ethics committee)
Record Dates: First submitted 2018-11-19; First posted 2018-11-28 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2020-09

CONDITIONS: Diabetic Neuropathy
Keywords: acupuncture; peripheral neuropathy; diabetes mellitus type II; neurophysiology; nerve conduction velocity
MeSH Terms: conditions — Diabetic Neuropathies; Peripheral Nervous System Diseases; Diabetes Mellitus, Type 2 | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: multicenter, open label, randomized
Masking Description: The statistician will be blinded to the study intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupuncture plus routine care (Experimental): 12 session of semistandardized acupuncture together with pharmacological routine care
  Interventions: Procedure: acupuncture; Drug: routine care
- routine care alone (Active Comparator): pharmacological routine care (antidepressants, anticonvulsants, opioids, nonsteroidal antiinflammatory drugs)
  Interventions: Drug: routine care

INTERVENTIONS:
Procedure: acupuncture — semistandardized selection of acupuncture points according to the clinical presentation of diabetic peripheral neuropathy (DPN) symptoms; 12 treatments over 8 weeks
  Arms: acupuncture plus routine care
Drug: routine care — pharmacological routine care (antidepressants, anticonvulsants, opioids, nonsteroidal antiinflammatory drugs)

SUMMARY:
Multicentric,randomized, two-armed confirmatory trial on the effectiveness of acupuncture in patients with symptomatic peripheral diabetic neuropathy compared to routine care.

DETAILED DESCRIPTION:
The study will investigate the effect of a series of acupuncture treatments on subdimensions of neuropathic symptoms, such as pain, tingling and numbness. Neurophysiological testing of the affected nerves are incorporated into the study as a possible morphological correlate of functional and clinical findings.

ELIGIBILITY:
Inclusion Criteria, among others:

* Diagnosis of diabetic peripheral neuropathy in diabetes mellitus Type 2
* Males and females aged >18yrs < 70yrs
* Minimum overall complaints of minimum 40mm on a visual analogue scale (VAS)
* Completed titration of pain medication against diabetic peripheral neuropathy
* Pathological nerve conduction velocity and amplitude of N. suralis ( <42meter/second and or < 6 mikroVolt)

Exclusion Criteria, among others:

* Very severe diabetic peripheral neuropathy with muscular weakness of proximal leg muscles
* Neuropathy due to other reasons such as borrelia infection, HIV, hereditary, alcohol toxic, or related to history of neurotoxic drugs.
* Severe peripheral artery disease Fontaine stage IV
* Ulcers or gangrenous lesions of the feet

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-03-02 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue Scale (VAS) general complaints and pain | 8 weeks
  Visual analogue Scale 100mm- ranging from 0mm no symptoms/ pain to 100mm worst imaginable symptoms or pain

SECONDARY OUTCOMES:
neuropathic pain symptom inventory (NPSI ) | average of last 24h at baseline, 8, 16, 24 weeks
  neuropathic pain symptom inventory- subdimensions of neuropathic pain are assessed in 10 of 11 Point numeric rating scales(NRS)
-diabetic peripheral neuropathic pain Impact measure (DPNPI) | average of last week at baseline, 8, 16, 24 weeks
  disease- specific Quality of Life- max sum score of 95; the higher the sum-score the higher the interference of diabetic peripheral neuropathy with activities of daily living.
Short-Form -12 (SF-12) | baseline , 8 weeks
  12 item Quality of Life- Questionnaire - different scores for subdimensions of daily living
pain perception Scale (SES german) | latest average at 8, 16, 24 weeks
  emotional component of pain -scale- max sum score of 96- the higher the score the higher the negative emotional burden of pain experience.
Patient global impression of Change (PGIC) | 8, 16 and 24 weeks
  Scale from 1= very much improved to 7= very much worse
neurophysiological assessment of Nervus Suralis nerve conduction velocity | baseline, 8,16 and 24 weeks
  measurements of nerve conduction velocity in meter per seconds (m/s)with device DPNCheck® Neurometrix®
neurophysiological assessment of Nervus Suralis height of amplitude of action potential | baseline, 8,16 and 24 weeks
  height of amplitude of action potential of N. suralis in mikroVolt (µV) with device "DPNCheck®" from Neurometrix®

CONTACTS AND LOCATIONS:
Overall Officials: Benno Brinkhaus, MD, PhD, Principal Investigator — Charite University, Berlin, Germany
Locations (2):
- Germany (2):
  - Charité Universitätsmedizin Campus Mitte, Berlin
  - Praxis für TCM am UKE, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weidenhammer W, Streng A, Linde K, Hoppe A, Melchart D. Acupuncture for chronic pain within the research program of 10 German Health Insurance Funds--basic results from an observational study. Complement Ther Med. 2007 Dec;15(4):238-46. doi: 10.1016/j.ctim.2006.09.005. Epub 2006 Oct 30. PMID 18054725
- [Background] Schroder S, Liepert J, Remppis A, Greten JH. Acupuncture treatment improves nerve conduction in peripheral neuropathy. Eur J Neurol. 2007 Mar;14(3):276-81. doi: 10.1111/j.1468-1331.2006.01632.x. PMID 17355547
- [Background] Witt CM, Pach D, Brinkhaus B, Wruck K, Tag B, Mank S, Willich SN. Safety of acupuncture: results of a prospective observational study with 229,230 patients and introduction of a medical information and consent form. Forsch Komplementmed. 2009 Apr;16(2):91-7. doi: 10.1159/000209315. Epub 2009 Apr 9. PMID 19420954
- [Derived] Bolster M, Dietzel J, Habermann IV, Horder S, Brinkhaus B, Stockigt B. Patients' experiences with acupuncture for diabetic polyneuropathy as part of a randomized controlled trial (ACUDPN) - a qualitative study. BMC Complement Med Ther. 2025 Sep 1;25(1):317. doi: 10.1186/s12906-025-05064-w. PMID 40890741
- [Derived] Dietzel J, Horder S, Habermann IV, Meyer-Hamme G, Hahn K, Ortiz M, Roll S, Linde K, Irnich D, Hammes M, Nogel R, Wullinger M, Wortman V, Hummelsberger J, Willich SN, Schroder S, Brinkhaus B. Acupuncture in diabetic peripheral neuropathy-protocol for the randomized, multicenter ACUDPN trial. Trials. 2021 Feb 26;22(1):164. doi: 10.1186/s13063-021-05110-1. PMID 33637134